CLINICAL TRIAL: NCT06625060
Title: A Multicentre, Randomised, Double-blind, Placebo-controlled, Dose Escalation and Dose Finding Phase II Study to Evaluate the Safety and Efficacy of IPN10200 in the Prevention of Episodic or Chronic Migraine in Adults
Brief Title: A Study to Evaluate IPN10200 Safety and Efficacy in the Prevention of Episodic or Chronic Migraine in Adults
Acronym: MERANTI
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLIN-10200-454
Record Dates: First submitted 2024-10-01; First posted 2024-10-03 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Episodic Migraine; Chronic Migraine

STUDY DESIGN:
Intervention Model Description: Model Description
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Masking Description
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (10):
- Step 1 - Cohort 1- IPN10200 (Experimental): Participants will receive IPN10200 dose A through injections at Day 1.
  Interventions: Biological: IPN10200
- Step 1 - Cohort 1 - Placebo (Placebo Comparator): Participants will receive placebo through injections at Day 1.
  Interventions: Other: Placebo
- Step 1 - Cohort 2 - IPN10200 (Experimental): Participants will receive IPN10200 dose B through injections at Day 1.
  Interventions: Biological: IPN10200
- Step 1 - Cohort 2 - Placebo (Placebo Comparator): Participants will receive placebo through injections at Day 1.
  Interventions: Other: Placebo
- Step 2- EM group IPN10200 Dose A (Experimental): Dose A will be administered to the participants in a single treatment cycle.
  Interventions: Biological: IPN10200 dose A
- Step 2- EM group IPN10200 Dose B (Experimental): Dose B will be administered to the participants in a single treatment cycle
  Interventions: Biological: IPN10200 dose B
- Step 2- EM group placebo (Placebo Comparator): Placebo will be administered to the participants in a single treatment cycle
  Interventions: Other: Placebo
- Step 2- CM group IPN10200 Dose A (Experimental): Dose A will be administered to the participants in a single treatment cycle
  Interventions: Biological: IPN10200 dose A
- Step 2- CM group IPN10200 Dose B (Experimental): Dose B will be administered to the participants in a single treatment cycle
  Interventions: Biological: IPN10200 dose B
- Step 2- CM group placebo (Placebo Comparator): Placebo will be administered to the participants in a single treatment cycle
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: IPN10200 — Lyophilised powder
  Arms: Step 1 - Cohort 1- IPN10200; Step 1 - Cohort 2 - IPN10200
Other: Placebo — Excipients without active substance, Lyophilised powder
  Arms: Step 1 - Cohort 1 - Placebo; Step 1 - Cohort 2 - Placebo; Step 2- CM group placebo; Step 2- EM group placebo
Biological: IPN10200 dose A — Lyophilised powder
  Arms: Step 2- CM group IPN10200 Dose A; Step 2- EM group IPN10200 Dose A
Biological: IPN10200 dose B — Lyophilised powder
  Arms: Step 2- CM group IPN10200 Dose B; Step 2- EM group IPN10200 Dose B

SUMMARY:
A migraine is a headache with severe throbbing pain or a pulsating sensation, usually on one side of the head. It is often accompanied by feeling or being sick and a sensitivity to bright lights and sound. Migraines are caused by a series of events when the brain gets stimulated or activated, which causes the release of chemicals that cause pain. IPN10200 is a medication that stops the release of these chemical messengers.

Participants with episodic migraine (EM) or chronic migraine (CM) will be included in both Step 1 and Step 2. "Headache days" are when participants experience headaches that meet the criteria for a migraine or a headache without the additional migraine-specific symptoms. "Migraine days" occur when the headache displays clear migraine characteristics.

This study aims to determine:

* The safety and efficacy of injecting IPN10200 directly into the muscles of the head and neck to prevent EM and CM,
* The right amount (dose) of IPN10200 to inject at each point,
* The total amount (dose) of IPN10200 that provides the best balance between safety and efficacy preventing migraines.

Participants will need to complete a daily electronic migraine Diary (eDiary) and questionnaires throughout the study. The total study duration for a participant will be up to 44 weeks.

DETAILED DESCRIPTION:
The study will consist of 3 periods:

1. A 'screening period' to assess whether the participant can take part in the study.
2. Step 1 is divided in two cohorts. The study will assess sequentially the safety of two doses of IPN10200, a lower dose in the cohort 1 and a higher dose in cohort 2. Participants will be administered with the study drug or placebo. The treatment is injected in muscles of the head, face and neck. The safety of participants is monitored throughout the 36 weeks at each cohort.
3. Step 2: In this step, new eligible participants will be divided into two groups based on their diagnosis (EM or CM). These groups will then be randomly assigned to one of three intervention groups: Dose A, Dose B, or a placebo. The intervention will be given in a series of injections in muscles of the head, face and neck. Participants will be monitored for both efficacy and safety until they complete the Week 36 visit (the end of study).

ELIGIBILITY:
Inclusion Criteria:

1. Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the ICF. Participant has provided written informed consent and signed privacy/data protection documentation;
2. Male or female ≥18 to 80 years of age at the time of signing the informed consent;
3. Diagnosis of either EM or CM, per ICHD-3 criteria, for at least 12 months prior to the screening visit;
4. Diagnosis of migraine at ≤50 years of age;
5. Participants in the EM group: History of EM diagnosis and headache frequency (i.e. migraine and non-migraine headache): ≤14 headache days in the 4 weeks prior to randomisation on study Day 1 based on information recorded in the eDiary; migraine frequency: ≥6 migraine days in the 4 weeks prior to randomisation on study Day 1 based on information recorded in the eDiary;
6. Participants in the CM group: History of CM diagnosis and headache frequency (i.e. migraine and non-migraine headache): ≥15 headache days in the 4 weeks prior to randomisation on study Day 1 based on information recorded in the eDiary; migraine frequency: ≥8 migraine days in the 4 weeks prior to randomisation on study Day 1 based on information recorded in the eDiary;
7. Participant with a history of use of at least one preventive treatment for migraine.

Exclusion Criteria:

1. History or current diagnosis of migraine with brainstem aura, retinal migraine, complications of migraine, tension-type headache, trigeminal autonomic cephalalgias, hypnic headache, hemicrania continua or new daily persistent headache;
2. Headache attributed to another disorder (e.g. secondary headaches), except medication overuse headache (MOH);
3. Current uncontrolled psychiatric or psychological condition, or one that could confound assessment of headaches/migraines or interfere with study participation;
4. Risk of self-harm or harm to others as evidenced by past suicidal behaviour or endorsing items 3, 4, or 5 on the C-SSRS at screening or Day 1.
5. Participants presenting with a swallowing disorder of any origin which might be exacerbated by botulinum toxin treatment, such as:

   - Grade 3 or 4 on the Dysphagia Severity Scale (severe dysphagia) with swallowing difficulties and requiring a change in diet.
6. Clinically relevant skin condition or infection that could interfere with injection of study intervention;
7. Participant has any medical condition or situation that would make them unsuitable for participation in the study;
8. Participant receiving more than one allowable concomitant migraine preventive treatment;
9. Known history of an inadequate response to >4 medications prescribed for the prevention of migraine (2 of which have different mechanisms of action to botulinum toxin);
10. Use of any of the following medications in the specified timeframe prior to the screening visit:

    * Botulinum toxin for migraine within 24 weeks (or for any other medical/aesthetic reason within 16 weeks);
    * Prior use of mAbs blocking CGRP pathway within 12 weeks for preventative treatment of migraine
    * Prior use of oral CGRP receptor antagonist (gepants) for preventative treatment of migraine within 2 weeks;
    * Anaesthetic or steroid injection in any region targeted for treatment with study medication within 4 weeks;
    * Use of cannabidiol or other types of cannabinoids within 30 days;
    * Use of medical device to treat migraine within 4 weeks (e.g. non-invasive neuromodulation therapies such as nerve stimulation (gammaCore), transcranial magnetic stimulation (cephaly), external trigeminal nerve stimulation, transcutaneous electrical nerve stimulation and peripheral neuroelectrical stimulation);
    * Use of other intervention to treat migraine that is assessed to interfere with study evaluations within 4 weeks (e.g. acupuncture in the head and neck region, cranial traction, nociceptive trigeminal inhibition, occipital nerve block treatments and dental splints for headache);
    * Use of opioids or barbiturates for more than 2 days/month within the last 4 weeks.
11. Concurrent participation in another interventional clinical study (or within specified timeframe according to national or local legislation or requirements);
12. Diagnosis of other significant pain disorders that could confound the assessment of headaches/migraines or interfere with study participation, including but not limited to chronic pain disorders such as fibromyalgia, chronic low back pain and complex regional pain syndrome;
13. Pregnant women, nursing women, premenopausal women, or WOCBP (i.e. not surgically sterile or 1 year postmenopausal) not willing to practice an acceptable contraceptive method, at the beginning of the study and for a minimum of 12 weeks following the administration of study treatment;
14. Male subjects who are not vasectomised and who have female partners of childbearing potential and are not willing to use condoms with spermicide for a minimum of 12 weeks following the initial double-blind administration of the treatment;
15. History of alcohol or drug abuse within 5 years of the screening visit (excluding medication overuse for headache);
16. Body mass index (BMI) ≥35 kg/m² at the screening visit;
17. Known clinically significant hypersensitivity to any of the study drugs, excipients or materials used to administer the study drug;
18. Patients who, in the clinician's judgment, are actively suicidal, and therefore, deemed to be at significant risk for suicide.
19. A diagnosis of a neuromuscular disorder or respiratory disorder, such as myasthenia gravis, Lambert-Eaton syndrome or amyotrophic lateral sclerosis that in the opinion of the investigator would compromise the safety of the study participant.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 641 (Estimated)
Dates: Start 2024-10-10 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-06-15 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants experiencing any Adverse Event (AEs) including treatment emergent adverse events (TEAEs), serious adverse events (SAEs), adverse event of special interest (AESI) and AE leading to treatment discontinuation | For step 1: From baseline until end of study at Week 36
  An Adverse event (AE) is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. TEAE is an AE for which the start date is on or after the date that the intervention began.
Percentage of Participants with clinically significant changes from baseline in Laboratory Parameters | For step 1: At all timepoints post injection until Week 36
  Clinically significant change in laboratory parameters will be reported. The clinical significance will graded by the investigator.
Percentage of Participants With Clinically Significant Changes from baseline in Vital Signs | For step 1: At all timepoints post injection until Week 36
  Clinically significant changes in vital signs will be reported. The clinical significance will be graded by the investigator.
Percentage of participants with clinically significant change from baseline in facial examination | For step 1: At all timepoints post injection until Week 36
  Clinically significant changes in facial examination and focused neurological/physical examinations will be reported. The clinical significance will be graded by the investigator.
Percentage of participants with clinically significant change from baseline in 12-lead Electrocardiogram (ECG) readings | For step 1: At all timepoints post injection until Week 36
Treatment-emergence of suicidal ideation/suicidal behaviour | For step 1: At all timepoints post injection until Week 36
  It will be assessed by the Columbia-Suicide Severity Rating Scale (C-SSRS) questionnaire that consists of 2 subscales:
  1. Ideation severity subscale: questions answered yes/no, severity of ideation scored 1-5 with 5 being most severe
  2. Intensity of ideation subscale : scores range from 2-25 with higher scores indicating more severe intensity of ideation.
Percentage of participants with Binding antibodies to IPN10200 | For step 1: At baseline, Week 4, Week 12 and Week 36.
Percentage of participants with neutralising antibodies to IPN10200 | For step 1: At baseline, Week 4, Week 12 and Week 36.
Change from baseline in the number of Monthly migraine days (MMD)s | For step 2: At Week 12 (Weeks 9-12).

SECONDARY OUTCOMES:
Change from baseline in the number of MMD | For Step 1 and step 2: From Week 1 to Week 36.
Change from baseline in the number of Monthly Headache Days (MHD) | For Step 1 and step 2: From Week 1 to Week 36
Change from baseline in the number of moderate/severe MHD | For Step 1 and step 2: From Week 1 to Week 36
Migraine prevention response | For Step 1 and step 2: From Week 1 to Week 36
  Migraine prevention response is assessed using two thresholds: by a reduction from baseline of either ≥50% or ≥75% in MMD
Headache prevention response | For Step 1 and step 2: From Week 1 to Week 36.
  Assessed using two thresholds: by a reduction from baseline of either ≥50% or ≥ 75% in MHD
Change from baseline in the number of days per 4 week period of acute medication use for migraine relief. | For Step 1 and step 2: From Week 1 to Week 36.
  An acute medication use day is defined as any day on which a participant reports, per eDiary, the intake of allowed medication(s) for the acute treatment of migraine.
The use of acute migraine medication (yes or no) | For Step 1 and step 2: From Week 1 to Week 36.
  The use of acute migraine medication will be recorded in the daily eDiary.
Percentage of participants with Binding antibodies to IPN10200 | For step 2 : At baseline, Week 4, Week 12 , Week 24 and Week 36.
Percentage of participants with neutralising antibodies to IPN10200 | For step 2 : At baseline, Week 4, Week 12 , Week 24 and Week 36.

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (166):
- United States (71):
  - Central Research Associates, Birmingham, Alabama
  - Rehabilitation & Neurological Services, LLC, Huntsville, Alabama
  - MD First Research - Chandler - Neurology, Chandler, Arizona
  - MD First Research - Chandler, Chandler, Arizona
  - Baptist Health Center for Clinical Research, Little Rock, Arkansas
  - Axiom Research, LLC, Apple Valley, California
  - Profound Research. LLC - NCSC, Carlsbad, California
  - M3Wake -PRI Encino, Encino, California
  - WR-PRI Encino, Encino, California
  - Neuro-Pain Medical Center, Fresno, California
  - Fullerton Neurological Center - Neurology, Fullerton, California
  - Neurology Center of North Orange County, Fullerton, California
  - University of California, Irvine - Department of Neurology, Irvine, California
  - Kaizen Brain Center, La Jolla, California
  - Pharmacology Research Institute (PRI), Los Alamitos, California
  - Pharmacology Research Institute (PRI) - Los Alamitos/Long Beach, Newport Beach, California
  - Profound Research, LLC, Pasadena, California
  - Acclaim Clinical Research - Internal Medicine, San Diego, California
  - Clinical Trials Management LLC, Thousand Oaks, California
  - Alliance Clinical West Hills (Focus Clinical Research), West Hills, California
  - Advanced Neuroscience Research Center, LLC, Fort Collins, Colorado
  - Advanced Neuroscience Research Center, LLC - Neurology, Fort Collins, Colorado
  - New England Institute for Neurology and Headache (NEINH)/Medical Practice, Stamford, Connecticut
  - Neurology Offices, Boca Raton, Florida
  - AGA Clinical Trials, Hialeah, Florida
  - M3 Wake Research/MSRA, LLC, Lake City, Florida
  - M3 Wake Research/MSRA,LLC, Lake City, Florida
  - Renstar Medical Research, Ocala, Florida
  - Clinical Neuroscience Solutions, Inc., Orlando, Florida
  - Emerald Coast Center For Neurological Disorders, Pensacola, Florida
  - Conquest Research, Winter Park, Florida
  - NeuroTrials Research, Inc., Atlanta, Georgia
  - Crescent City Headache and Neurology Center, LLC, Chalmette, Louisiana
  - Ochsner Health Center - Covington, Covington, Louisiana
  - DelRicht Research, New Orleans, Louisiana
  - DelRicht Research at Touro Medical Center, New Orleans, Louisiana
  - LSU Healthcare Network Orthopedic & Sports Medicine, New Orleans, Louisiana
  - MedStar Neurosciences and Rehabilitation Research Network, Baltimore, Maryland
  - MedStar Neurosciences and Rehabilitation, Baltimore, Maryland
  - MedStar Franklin Square Hospital Center, Baltimore, Maryland
  - Medstar Franklin Square Medical Center, Baltimore, Maryland
  - Neurology Center of NE,PC - Neurology, Foxborough, Massachusetts
  - MedVadis Research, Waltham, Massachusetts
  - Mass Institute of Clinical Research, Westborough, Massachusetts
  - Michigan Head Pain & Neurological Institute - Neurology/Pain, Ann Arbor, Michigan
  - Michigan Head Pain & Neurological Institute, Ann Arbor, Michigan
  - Michigan Center of Medical Research, Grand Blanc, Michigan
  - Minneapolis Clinic-Neurology, Burnsville, Minnesota
  - Papillion Research Center/Avacare, Papillion, Nebraska
  - Alliance Clinical Las Vegas (Excel Clinical Research) - Internal Medicine, Las Vegas, Nevada
  - Integrative Clinical Trials, LLC, Brooklyn, New York
  - Montefiore Medical Center: Headache Center, The Bronx, New York
  - Upstate Clinical Research Associates - Research Center, Williamsville, New York
  - Upstate Clinical Research Associates, Williamsville, New York
  - UC Gardner Neuroscience Institute, Cincinnati, Ohio
  - Neurology Diagnostics, Inc., Dayton, Ohio
  - Mount Carmel Health Systems, New Albany, Ohio
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Preferred Primary Care Physicians - Curry Hollow, Pittsburgh, Pennsylvania
  - Clinical Neuroscience Solutions, Inc - Memphis, Memphis, Tennessee
  - Clinical Neuroscience Solutions, Inc., Memphis, Tennessee
  - Zenos Clinical Research - Internal Medicine, Dallas, Texas
  - Lone Star Neurology, Frisco, Texas
  - Elevate Clinical Research - Houston, Houston, Texas
  - Javara Inc. - Houston, TX, Houston, Texas
  - Javara Inc. - New Caney, TX, New Caney, Texas
  - J. Lewis Research-Site Number:8400053, Salt Lake City, Utah
  - ChronicleBio, West Valley City, Utah
  - Puget Sound Neurology - Neurology, Tacoma, Washington
  - Marshall Health Clinical Research Center, Huntington, West Virginia
  - Frontier Clinical Research, LLC - Kingwood, Kingwood, West Virginia
- Australia (3):
  - The Alfred Hospital - Neurology, Melbourne
  - Western Health - Neurology & Stroke Services, Saint Albans
  - The Royal Melbourne Hospital - Neurology, Victoria Park
- Brazil (5):
  - Instituto de Neurologia de Curitiba, Paraná
  - Associação Hospitalar Moinhos de Vento, Rio Grande
  - A2Z Clinical, São Paulo
  - Hospital Alemao Oswaldo Cruz, São Paulo
  - Pseg Centro de Pesquisa Clínica S.A, São Paulo
- Canada (6):
  - CaRe Clinic - Calgary, Calgary
  - University of Calgary Foothills Campus, Calgary
  - Centre de Recherche Saint-Louis (Lévis) - Clinique Neuro-Lévis, Lévis
  - Centre de Recherche Saint-Louis (Quebec) - Clinique Médicale Saint-Louis, Québec
  - CaRe Clinic Red Deer, Red Deer
  - Bluewater Clinical Research Group Inc., Sarnia
- Czechia (7):
  - Pratia Brno s.r.o., Brno
  - NEUROHK s.r.o., Choceň
  - NeuropsychiatrieHK, s.r.o., Hradec Králové
  - Fakultni nemocnice Ostrava - Neurologicka klinika, Ostrava
  - Pratia Pardubice a.s., Pardubice
  - AXON clinical, Prague
  - DADO MEDICAL s.r.o., Prague
- France (5):
  - CHU Amiens Sud-Centre Rech Clinique, Amiens
  - Centre Hospitalier Regional Universtaire De Clermont-Ferrand - Neurologie, Clermont-Ferrand
  - CHU de Nantes - HÃ´pital Laennec - Neurology, Nantes
  - CHU Nimes - Hôpital Caremeau - Service de Neurologie, Nîmes
  - Assistance Publique-Hopitaux de Paris (AP-HP) - Unite de Recherche Clinique Saint-Louis Lariboisere-Ferd Widal, Paris
- Georgia (6):
  - Ltd "Health", Batumi
  - "Pineo Medical Ecosystem" LTD, Tbilisi
  - LTD "Israel-Georgian Medical Research Clinic Healthycore", Tbilisi
  - LTD "Multiprofile Clinic Consilium Medulla", Tbilisi
  - LTD New Hospitals - Neurology, Tbilisi
  - Ltd. S.Khechinashvili University Clinic, Tbilisi
- Germany (10):
  - Charite - Universitaetsmedizin Berlin - Neurology, Berlin
  - FutureMeds Berlin (emovis), Berlin
  - Universitaetsklinikum Carl Gustav Carus an der Technischen Universitaet Dresden - UniversitaetsSchmerzCentrum - USC, Dresden
  - Universitätsklinikum Essen (AöR), Essen
  - Kopfschmerzzentrum Frankfurt, Frankfurt
  - Praxis Dr. Oehlwein, Gera
  - Schmerz- und Palliativzentrum Goeppingen, Göppingen
  - Universitaetsmedizin Greifswald, Greifswald
  - Neurologisch-verhaltensmedizinische Schmerzklinik Kiel, Kiel
  - NeuroPoint, Ulm
- Japan (11):
  - Ikeda Neurosurgical Clinic - Neurosurgery, Fukuoka
  - DOI Internal Medicine/Neurology Clinic, Hiroshima
  - Konankai Konan Medical Center - Neurology, Hyōgo
  - Tanaka Neurosurgery & Headache Clinic, Kagoshima
  - Ishikawa Clinic, Kyoto
  - Sendai Zutsu No-Shinkei Clinic - Neurology, Miyagi
  - Tominaga Clinic - Neurology, Osaka
  - Japanese Red Cross Shizuoka Hospital - Neurology, Shizuoka
  - Iwata Neurosurgery Clinic, Tokyo
  - Kitasato University Kitasato Institute Hospital - Urology - Neurology, Tokyo
  - Nagamitsu Clinic - Neurology, Yamaguchi
- New Zealand (7):
  - Optimal Clinical Trials, Auckland
  - New Zealand Brain Research Institute at University of Otago, Christchurch
  - Optimal Clinical Trials - Christchurch, Christchurch
  - Pacific Clinical Research Network (PCRN) - Christchurch, Christchurch
  - Pacific Clinical Research Network (PCRN) - Tasman, Nelson
  - Pacific Clinical Research Network (PCRN) - Auckland, Takapuna
  - Lakeland Clinical Trials Wellington, Upper Hutt
- Poland (17):
  - Synexus Polska Sp. z o.o., Częstochowa
  - Silmedic sp. z o.o., Katowice
  - Synexus Katowice, Katowice
  - Uniwersyteckie Centrum Kliniczne im. prof. K. Gibinskiego Slaskiego Uniwersytetu Medycznego w Katowicach, Katowice
  - Centrum Medyczne PROMED, Krakow
  - CM Linden, Krakow
  - FutureMeds Krakow, Krakow
  - Specjalistyczne Gabinety Sp. z o.o., Krakow
  - FutureMeds Lodz, Lodz
  - Instytut Zdrowia Dr Boczarska-Jedynak Sp. z o.o. S.K., Oświęcim
  - Synexus Polska Sp. z o.o. - Oddzial w Gdyni, Pomorskie
  - Velocity Nova Sp. z o.o - Velocity Pulawy, Puławy
  - ETG Siedlce, Siedlce
  - Centrum Leczenia Zaburzen Pamieci i Neuroobrazowania Affidea, Warsaw
  - City Clinic Research Sp. z o.o., Warsaw
  - ETG Neuroscience Sp. z o.o., Warsaw
  - MIGRE Polskie Centrum Leczenia Migreny Anna Gryglas-Dworak, Wroclaw
- South Korea (7):
  - Hallym University Dongtan Sacred Heart Hospital - Neurology, Gyeonggi-do
  - Inje University Ilsan Paik Hospital - Allergology, Gyeonggi-do
  - Ewha Womans University Seoul Hospital - Neurology, Seoul
  - Kangbuk Samsung Hospital - Neurology, Seoul
  - Nowon Eulji Medical Center, Eulji University - Neurology, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
- Spain (7):
  - Hospital Clinic de Barcelona - Neurología, Barcelona
  - Hospital Universitario Vall d'Hebron - Enfermedades Infecciosas, Barcelona
  - FutureMeds Spain Cádiz, Cadiz
  - FutureMeds Madrid, Madrid
  - Hospital Universitario MarquÃ©s de Valdecilla - Neurologia, Santander
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Clinico Universitario de Valladolid - Gastroenterology, Valladolid
- United Kingdom (4):
  - Royal Devon And Exeter Hospital - Neurology, Exeter
  - Hull University Teaching Hospitals NHS Trust - Hull Royal Infirmary, Hull
  - Walton Centre For Neurology And Neurosurgery, Liverpool
  - King's College Hospital, London

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, annotated case report form, statistical analysis plan, and dataset specifications.
  Patient level data will be anonymized and study documents will be redacted to protect the privacy of study participants.
Time Frame: Where applicable, data from eligible studies are available 6 months after the studied medicine and indication have been approved in the US and/or EU.
Access Criteria: Further details on Ipsen's sharing criteria and process for sharing are available here (https://www.ipsen.com/science/clinical-trials/clinical-data-transparency/).
URL: https://www.ipsen.com/science/clinical-trials/clinical-data-transparency/